CLINICAL TRIAL: NCT05647720
Title: Effect of Maxillary Third Molar Extraction vs Non-extraction on Distalization of First Molars in a Group of Adolescent Patients Using Infra-Zygomatic Gear Distalizer: A Randomized Clinical Trial
Brief Title: Effect of Maxillary Third Molar Extraction vs. Non-extraction on Distalization of First Molars in a Group of Adolescent Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Nadeen Hafez, Principal investigator, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUE.REC(14)/7-2019
Record Dates: First submitted 2022-11-25; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Class II Malocclusion
Keywords: Infra-zygomatic mini-implant; Distalization; Infra-zygomatic crest; Digital models; molar tipping
MeSH Terms: conditions — Overbite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Only the outcome assessors will be blind. The patients name will be sealed from the pre- and post-radiographs and study models. Then two assessors will carry out, blindly and independently, the measurements and analysis of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Third molar extraction group (Experimental): After surgical extraction of unerupted upper third molars, the maxillary first molars were distalized using the infra-zygomatic gear distalizer, which is anchored to infra-zygomatic mini-implants inserted in the infra-zygomatic crest.
  Interventions: Procedure: Distalization combined with upper third molars extraction
- Third molar presence group (Experimental): Without extraction of unerupted upper third molars, the maxillary first molars were distalized using the infra-zygomatic gear distalizer, which is anchored to infra-zygomatic mini-implants inserted in the infra-zygomatic crest.
  Interventions: Procedure: Distalization without upper third molars extraction

INTERVENTIONS:
Procedure: Distalization combined with upper third molars extraction — After surgical extraction of unerupted upper third molars, the maxillary first molars were distalized using a labial bow with two soldered crimpable hooks distal to the upper lateral incisors. The labial bow fitted in the flying tube of the upper first molar bands. It was anchored bilaterally to the infra-zygomatic mini-implant by closed coil spring that applied a force of 300gm on each side
  Arms: Third molar extraction group
Procedure: Distalization without upper third molars extraction — The maxillary first molars were distalized , without extracting upper third molars, using a labial bow with two soldered crimpable hooks distal to the upper lateral incisors. The labial bow fitted in the flying tube of the upper first molar bands. It was anchored bilaterally to the infra-zygomatic mini-implant by closed coil spring that applied a force of 300gm on each side
  Arms: Third molar presence group

SUMMARY:
There is a scarcity in literature regarding the influence of maxillary third molar on distalization . This study aimed to compare the influence of unerupted maxillary third molars and their extraction on the bilateral distalization of upper first molars using the infra-zygomatic gear distalizer

DETAILED DESCRIPTION:
Maxillary molar distalization is one of the non-extraction modalities for treating class II malocclusion. When distalizing maxillary molars In adults, it is not a problem to extract fully erupted third molars, and it may even be suggested that the extraction site may accommodate distalization. On the contrary, adolescents usually have unerupted third molars with partially formed roots, rendering the surgical extraction more difficult and traumatic. The necessity of surgically extracting upper third molar buds before distalization remains questionable. Therefore, this study was conducted to three-dimensionally assess the impact of maxillary third molar presence on distalizing maxillary molars in adolescent patients having Class II malocclusion.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent patients aged 16-19 years
* skeletal Class I
* bilateral Class II molar relationship. defined by at least an end-to-end molar relationship.
* normal vertical growth pattern.
* full permanent dentition with unerupted upper third molars.

Exclusion Criteria:

* skeletal Class II or Class III relationship.
* past orthodontic treatment.
* poor oral hygiene.
* Increased vertical dimension.

Ages: 16 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2021-02-28 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
distalization amount of maxillary firs molars at the crown and root levels | From pre to post distalization (an average of 8 months)
  Anteroposterior changes in the position of maxillary first molars assessed on digitized models and cone beam computed tomography (CBCT) taken for each patient before and after distalization. Measurements were done by identifying landmarks, reference lines, and planes(measured in mm)

SECONDARY OUTCOMES:
Rate of maxillary first molar Distalization | From pre- to post-distalization (an average of 8 months)
  Incremental changes in the antero-posterior position of maxillary first molars assessed on digitized models taken for each patient before and after distalization and in each follow up visit. Measurements were done by identifying landmarks, reference lines, and planes (measured in mm)
Tipping of maxillary first molar | From pre- to post-distalization (an average of 8 months)
  Angular changes of maxillary first molar assessed on cone beam computed tomography (CBCT) taken for each patient before and after distalization. Measurements were done by identifying landmarks, reference lines, and planes(measurement of the angles in degrees).
Vertical position of maxillary first molar | From pre- to post-distalization (an average of 8 months)
  vertical positional changes of maxillary first molar assessed on cone beam computed tomography (CBCT) taken for each patient before and after distalization. Measurements were done by identifying landmarks, reference lines, and planes (measured in mm)
Inter molar width | From pre- to post-distalization (an average of 8 months)
  Changes in the transvers distance between the right and left upper first molars assessed on digitized models taken for each patient before and after distalization. Measurements were done by identifying landmarks, reference lines, and planes (measured in mm)
Molar rotation | From pre- to post-distalization (an average of 8 months)
  Study models that are taken pre and post retraction (then digitalized) will be used to assess the rotation of the maxillary first molars in relation to a reference line (measurement of the angles in degrees)
Tipping of maxillary second molar | From pre- to post-distalization (an average of 8 months)
  Angular changes of maxillary second molar assessed on cone beam computed tomography (CBCT) taken for each patient before and after distalization. Measurements were done by identifying landmarks, reference lines, and planes. (measured in of in degrees)
Tipping of maxillary third molar | From pre- to post-distalization (an average of 8 months)
  Angular changes of maxillary third molar assessed on cone beam computed tomography (CBCT) taken for each patient before and after distalization. Measurements were done by identifying landmarks, reference lines, and planes (measurement of the angles in degrees)
Vertical position of maxillary third molar | From pre- to post-distalization (an average of 8 months)
  Vertical positional changes of maxillary third molar assessed on cone beam computed (measured in mm)tomography (CBCT) taken for each patient before and after distalization. Measurements were done by identifying landmarks
  , reference lines, and planes (measured in mm)
Vertical position of upper incisors | From pre- to post-distalization (an average of 8 months)
  Vertical positional changes of upper incisors assessed on cone beam computed tomography (CBCT) taken for each patient before and after distalization. Measurements were done by identifying landmarks, reference lines, and planes (measured in mm)
Anteroposterior position of upper incisors | From pre- to post-distalization (an average of 8 months)
  Antero-posterior change in the anteroposterior position of upper incisors assessed on cone beam computed tomography (CBCT) taken for each patient before and after distalization. Measurements were done by identifying landmarks, reference lines, and planes (measured in mm)
upper incisors torque | From pre- to post-distalization (an average of 8 months)
  Angular changes of upper incisors assessed on cone beam computed tomography (CBCT) taken for each patient before and after distalization. Measurements were done by identifying landmarks, reference lines, and planes (measurement of the angles in degrees)
Anteroposterior changes of upper first and second premolars | From pre- to post-distalization (an average of 8 months)
  Antero-posterior change in the position of maxillary first and second premolars assessed on digitized models taken for each patient before and after distalization. Measurements were done by identifying landmarks, reference lines, and planes (measured in mm)

CONTACTS AND LOCATIONS:
Overall Officials: Yehya Mostafa, Professor and Chairman, Study Director — Future University in Egypt
Locations (1):
- Future University in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All collected participant data (IPD)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after publication

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT05647720/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT05647720/ICF_001.pdf